CLINICAL TRIAL: NCT05792488
Title: The Investigation of Different Guidance Methods to Facilitate Lifestyle Changes in Patients With NAFLD
Brief Title: Lifestyle Guidance Methods in NAFLD
Acronym: INDIANA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Mathieu Struyve, Principal Investigator, Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z-2022064
Record Dates: First submitted 2022-11-07; First posted 2023-03-31 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Doulas; Amyloid; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of care (Other)
  Interventions: Other: Standard of care
- Lifestyle coach (Experimental)
  Interventions: Behavioral: Coach
- App (Experimental)
  Interventions: Behavioral: App

INTERVENTIONS:
Behavioral: Coach — Coaching to a healthy lifestyle
  Arms: Lifestyle coach
Behavioral: App — The app will coach people to a healthy lifestyle
  Arms: App
Other: Standard of care — Patients will receive standardized lifestyle advice by their specialist
  Arms: Standard of care

SUMMARY:
To determine the efficiency of lifestyle modification (due to a dietitian or digital application) compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* NAFLD based in FibroScan measurements

Exclusion Criteria:

* excessive alcohol use
* other causes of liver disease
* secondary causes of liver steatosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
A change in liver fat | 1 year
  As measured by the controlled attenuation parameter in the intervention arms as compared to standard of care

CONTACTS AND LOCATIONS:
Overall Officials: Geert Robaeys, MD. PhD, Principal Investigator — Hasselt University
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided